CLINICAL TRIAL: NCT01917812
Title: mActive: A Blinded, Randomized mHealth Trial of Digital Activity Tracking and Smart Texting to Promote Physical Activity
Brief Title: mActive: A Blinded, Randomized mHealth Activity Trial
Acronym: mActive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: NA_00086400
Record Dates: First submitted 2013-08-01; First posted 2013-08-07 (Estimated); Results first posted 2016-01-05 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-02

CONDITIONS: Physical Activity
Keywords: physical activity; exercise; mHealth; smartphone; activity tracker; pedometer; text messaging; SMS
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Blinded Digital Activity Tracker (Placebo Comparator): Blinded Digital Activity Tracker = Group wears the tracker but is blinded to the numeric physical activity feedback information provided by the tracker.
  Interventions: Device: Digital Activity Tracker
- Unblinded Digital Activity Tracker / No Smart Text Messaging (Experimental): Unblinded Digital Activity Tracker = Group unblinded to the numeric physical activity feedback information provided by the digital activity tracker.
  No Smart Text Messaging = Group does not receive personalized, health coaching via "smart" text messages.
  Note that the study occurred over two study phases after the 1-week blinded run-in. In the first 2-week phase, participants were randomized to unblinded or blinded tracking. In the second 2-week phase, the unblinded participants were randomized to receive smart texts or no texts.
  Interventions: Device: Digital Activity Tracker
- Unblinded Digital Activity Tracker / Smart Text Messaging (Experimental): Unblinded Digital Activity Tracker = Group unblinded to the numeric physical activity feedback information provided by the digital activity tracker.
  Smart Text Messaging = Group receives personalized, health coaching via "smart" text messages.
  Note that the study occurred over two study phases after the 1-week blinded run-in. In the first 2-week phase, participants were randomized to unblinded or blinded tracking. In the second 2-week phase, the unblinded participants were randomized to receive smart texts or no texts.
  Interventions: Device: Digital Activity Tracker; Other: Smart Text Messaging

INTERVENTIONS:
Device: Digital Activity Tracker
  Other Names: Fitbug Orb
Other: Smart Text Messaging
  Arms: Unblinded Digital Activity Tracker / Smart Text Messaging

SUMMARY:
Despite their importance, health-related behaviors are hard to change. Among behaviors, physical activity is associated with protection from multiple diseases. People who are physically active have lower risk for heart disease, stroke, type 2 diabetes, depression, and some cancers with associated dose-dependent reductions in cardiovascular and all-cause mortality. However, most US adults do not meet CDC physical activity guidelines. Sedentary work behavior in industrialized nations is likely a contributor to this problem.

Current low-technology strategies for encouraging lifestyle change are disappointingly ineffective and are highly resource intensive. Systematic reviews of the literature show mixed evidence for using activity trackers (i.e., pedometers) and a limited body of evidence for text messaging in preventive health care. However, prior studies have not integrated digital activity tracking with mobile phone text messaging feedback.

Given 91% of adults in the United States now use a mobile phone, and 56% a smartphone, this represents a potentially widely applicable avenue for therapeutic intervention. There is growing interest in leveraging mobile health (mHealth) technologies to improve health behaviors in the general population. The investigators propose to conduct a blinded, randomized mHealth trial of digital activity tracking and smart texting to promote physical activity.

DETAILED DESCRIPTION:
Using an innovative, convenient, mHealth trial design, this pilot study aims to test the feasibility of a seamless model of information flow integrating digital activity tracker information with a mobile phone texting system to deliver a technology-enhanced intervention that does not require in-person follow-up.

The investigators hypothesize that:

1. individuals overestimate their physical activity, especially that done at work.
2. biofeedback from an activity tracker can increase physical activity via increasing self-awareness.
3. "smart" text message feedback can increase physical activity via personalizing health coaching.

Digitalized activity tracking will use the Fitbug Orb, which syncs via Bluetooth with one's smartphone. It is a display-free triaxial accelerometer, allowing one to blind participants to numeric feedback. Text messaging will use Reify Health's "smart" platform for personalized, interactive texting by an automated and repeatable algorithm. Texting will be informed by real-time activity information.

Potential advantages of the trial strategy include elimination of attendance at in-person sessions, personalization of health coaching, more continuous patient contact; inexpensive intervention, the ultimate ability to scale our intervention to larger target populations.

After initial pilot trial completion, additional study will include long-term physical activity follow-up of participants and focus groups.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to cardiology clinic
* Aged 18-69 years
* User of a compatible smartphone

Exclusion Criteria:

* Already using an activity tracker
* Preferred form of activity is not measured by an activity tracker(swimming, yoga, ice skating, stair master, or activities on wheels such as bicycling or rollerblading)
* Prohibited from normal activity due to wheelchair bound status, bed bound status, reliance on a cane/walker, activity-limiting pulmonary disease, activity-limiting angina, activity-limiting osteoarthritis, or other condition.
* 3 days or more of moderate or vigorous activity during leisure time for 30 minutes of more per day by International Physical Activity Questionnaire

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Blaha, MD, MPH, Study Director — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Result] Martin SS, Feldman DI, Blumenthal RS, Jones SR, Post WS, McKibben RA, Michos ED, Ndumele CE, Ratchford EV, Coresh J, Blaha MJ. mActive: A Randomized Clinical Trial of an Automated mHealth Intervention for Physical Activity Promotion. J Am Heart Assoc. 2015 Nov 9;4(11):e002239. doi: 10.1161/JAHA.115.002239. PMID 26553211
- See also: mActive: A Blinded, Randomized mHealth Trial Supporting Digital Tracking and Smart Texting for Promotion of Physical Activity. AHA EPI Scientific Sessions Presentation Slides. — http://my.americanheart.org/idc/groups/ahamah-public/@wcm/@sop/@scon/documents/downloadable/ucm_472545.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled outpatients at an academic cardiovascular prevention center (Johns Hopkins Ciccarone Center) in Baltimore, Maryland, USA from January 17 to May 20, 2014.
Groups:
- Blinded Digital Activity Tracker: Blinded Digital Activity Tracker = Group wears the tracker but is blinded to the numeric physical activity feedback information provided by the tracker.
  Blinded Digital Activity Tracker
- Unblinded Digital Activity Tracker / No Smart Text Messaging: Unblinded Digital Activity Tracker = Group unblinded to the numeric physical activity feedback information provided by the digital activity tracker.
  No Smart Text Messaging = Group does not receive personalized, health coaching via "smart" text messages.
  Unblinded Digital Activity Tracker
- Unblinded Digital Activity Tracker / Smart Text Messaging: Unblinded Digital Activity Tracker = Group unblinded to the numeric physical activity feedback information provided by the digital activity tracker.
  Smart Text Messaging = Group receives personalized, health coaching via "smart" text messages.
  Unblinded Digital Activity Tracker
  Smart Text Messaging
Period: Overall Study
Arm/Group | Blinded Digital Activity Tracker | Unblinded Digital Activity Tracker / No Smart Text Messaging | Unblinded Digital Activity Tracker / Smart Text Messaging
Started | 16 | 16 | 16
Completed | 15 | 16 | 16
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Unblinded Digital Activity Tracker / No Smart Text Messaging: Unblinded Digital Activity Tracker = Group unblinded to the numeric physical activity feedback information provided by the digital activity tracker.
  Unblinded Digital Activity Tracker
- Total: Total of all reporting groups
Arm/Group | Blinded Digital Activity Tracker | Unblinded Digital Activity Tracker / No Smart Text Messaging | Unblinded Digital Activity Tracker / Smart Text Messaging | Total
Number analyzed (Participants) | 16 | 16 | 16 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (7) | 58 (8) | 55 (8) | 58 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 8 | 22
  Male | 9 | 9 | 8 | 26
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 16 | 48

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily Step Count
Description: Note that the study occurred over two study phases after the 1-week blinded run-in. In the first 2-week phase, participants were randomized to unblinded or blinded tracking. In the second 2-week phase, the unblinded participants were randomized to receive smart texts or no texts.
Time Frame: Change from baseline mean daily step count at 3 weeks (end of unblinded digital activity tracker intervention)
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Blinded Digital Activity Tracker | Unblinded Digital Activity Tracker
Number analyzed (Participants) | 16 | 32
steps per day | -616 (2385) | 408 (2701)

2. Secondary Outcome: Mean Daily Activity Time
Description: as for outcome 1
Time Frame: Change from baseline mean daily activity time at 3 weeks (end of unblinded digital activity tracker intervention)
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Blinded Digital Activity Tracker | Unblinded Digital Activity Tracker
Number analyzed (Participants) | 16 | 32
minutes per day | -6 (26) | 2 (27)

3. Secondary Outcome: Mean Daily Aerobic Activity Time
Description: Defined as the time spent walking continuously for >10 minutes without breaking for more than a minute.
  Note that the study occurred over two study phases after the 1-week blinded run-in. In the first 2-week phase, participants were randomized to unblinded or blinded tracking. In the second 2-week phase, the unblinded participants were randomized to receive smart texts or no texts.
Time Frame: Change from baseline mean daily aerobic activity time at 3 weeks (end of unblinded digital activity tracker intervention)
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Blinded Digital Activity Tracker | Unblinded Digital Activity Tracker
Number analyzed (Participants) | 16 | 32
minutes per day | -11 (14) | -3 (12)

4. Primary Outcome: Mean Daily Step Count
Description: as for outcome 1
Time Frame: Change from 3 weeks mean daily step count at 5 weeks (end of smart text messaging intervention)
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Blinded Digital Activity Tracker | Unblinded Digital Activity Tracker | Unblinded Digital Activity Tracker / Smart Text Messaging
Number analyzed (Participants) | 16 | 16 | 16
steps per day | -1042 (2202) | -200 (1653) | 2334 (1714)

5. Secondary Outcome: Mean Daily Activity Time
Description: as for outcome 1
Time Frame: Change from 3 weeks mean daily activity time at 5 weeks (end of smart text messaging intervention)
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Blinded Digital Activity Tracker | Unblinded Digital Activity Tracker | Unblinded Digital Activity Tracker / Smart Text Messaging
Number analyzed (Participants) | 16 | 16 | 16
minutes per day | -8 (23) | 0 (17) | 21 (20)

6. Secondary Outcome: Mean Daily Aerobic Activity Time
Description: as for outcome 1
Time Frame: Change from 3 weeks mean daily aerobic activity time at 5 weeks (end of smart text messaging intervention)
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Blinded Digital Activity Tracker | Unblinded Digital Activity Tracker | Unblinded Digital Activity Tracker / Smart Text Messaging
Number analyzed (Participants) | 16 | 16 | 16
minutes per day | -3 (10) | -1 (8) | 13 (11)

ADVERSE EVENTS:
Arm/Group | Blinded Digital Activity Tracker | Unblinded Digital Activity Tracker / No Smart Text Messaging | Unblinded Digital Activity Tracker / Smart Text Messaging
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
Given its limited size and scope, mActive may be categorized as a pilot trial. As such, it is most appropriately interpreted as exploratory evidence to guide a definitive pivotal trial in the future.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No